CLINICAL TRIAL: NCT06594952
Title: Evaluation of Maternal Mental Health Following Ultrasonography Detection of Fetal Congenital Anomalies
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Areej Abdalrahman Khamees, Principal investigator, Assiut University
Other Study IDs: Maternal psychology on anomaly
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- minor anomalies group: pregnant women with minor fetal structural anomaly detected by ultrasound.
  Interventions: Other: Questionnaire and Physical Exam
- major anomalies group: pregnant women with major fetal structural anomaly detected by ultrasound
  Interventions: Other: Questionnaire and Physical Exam
- Control Group: Pregnant women with normal ultrasound.
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — Diagnosis of Anxiety using the state-trait anxiety inventory scale (STAI). Depression using Edinburgh Postnatal Depression Scale (EPDS)
  * Coping using the Brief Coping Scale
  * Socioeconomic using the Socioeconomic Scale of Egypt
  * Personality using the short-form Eysenck Personality Questionnaire-Revised (EPQ-R)
  * Behaviour using Impact of Erect Scale (IES-22)

SUMMARY:
The purpose of this study is to evaluate maternal mental health during antenatal and postnatal periods after Ultrasonography diagnosis of fetal anomalies.

DETAILED DESCRIPTION:
Fetal congenital anomalies are responsible for a great deal of abortions in desired pregnancies . In clinical practice, prenatal screening programs in 1st and 2nd trimester target both chromosomal and structural abnormalities. These congenital anomalies are classified as minor and major anomalies than may lead to death or stillbirth . Half of all anomalies are detectable during weeks 18-22 of pregnancy. Due to the advances occurring in Ultrasonography and screening paradigms, the rate of diagnosed anomalies is increasing dramatically which in turn leading to psychological distress in the pregnant mother. Receiving a diagnosis of fetal anomaly is a highly stressful and potentially traumatic event that can elicit immediate feelings of grief, loss, anger, depression, and anxiety. However, the foreknowledge of a fetal anomaly during pregnancy may enable the mother to prepare mentally resulting in reduced maternal stress after delivery. The American College of Medical Genetics recommends underscoring the importance of psychological assessment and substantive communication with parents facing a prenatal diagnosis of fetal anomaly. Despite the accessibility of establishing the significant symptoms of maternal psychological distress, the evidence on the definite nature of this distress in consideration to other life stressors and an accurate the prediction of women vulnerability in the critical period have not been clear yet due to many methodological issues. Identification of women at highest risk for poor adaptation to the diagnosis may allow for targeted psychological support services for those most vulnerable.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with confirmed pregnancy with viable fetus (whether singleton or multiple)
* Fetal anomaly should be diagnosed with ultrasonography (whether minor or major) after 12 weeks of gestational age

Exclusion Criteria:

- Women with history of psychiatric disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women receiving obstetric care at our tertiary perinatal care
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in anxiety scores between the study groups | 4 weeks
  using the state-trait anxiety inventory scale (STAI).

SECONDARY OUTCOMES:
Difference in Depression scores between the study groups | 4 weeks
  Depression using Edinburgh Postnatal Depression Scale (EPDS)

IPD SHARING:
Plan to Share IPD: No